CLINICAL TRIAL: NCT00171327
Title: Efficacy and Safety of Fluvastatin 80 mg or Valsartan 160 mg and Their Combination in Dyslipidemic Patients With Arterial Hypertension and Endothelial Dysfunction
Brief Title: Efficacy and Safety of Fluvastatin or Valsartan and Their Combination in Dyslipidemic Patients With Hypertension and Endothelial Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CXUO320BRU01
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension; Dyslipidemia
Keywords: arterial hypertension; dyslipidemia; valsartan; fluvastatin
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — Valsartan; Fluvastatin

INTERVENTIONS:
Drug: valsartan, fluvastatin

SUMMARY:
Patients with mild to moderate hypertension, dyslipidemia (imbalanced blood lipids) and decreased vascular dilatation, receiving a cholesterol lowering diet were given either valsartan or fluvastatin for 8 weeks. At week 8 all patients were administered a combination treatment with valsartan 160 mg and fluvastatin 80 mg.

ELIGIBILITY:
Inclusion Criteria:

* Arterial hypertension
* Dyslipidemia
* Cholesterol lowering diet

Exclusion Criteria:

* Constant antihypertensive treatment
* Diabetes mellitus
* Myocardial infarction or stroke in the previous 3 months

Other inclusion and exclusion criteria may apply

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2004-07; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in brachial artery flow-mediated vasodilation after 8 weeks
Percent change from baseline in brachial artery flow-mediated vasodilation after 16 weeks compared to 8 weeks

SECONDARY OUTCOMES:
Percent change from baseline in low density lipoprotein cholesterol, total cholesterol, and triglycerides
Evaluating blood pressure effect on endothelial function
Evaluating total cholesterol effect on endothelial function

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Principal Investigator — Novartis Pharmaceuticals
Locations (1):
- Novartis, Moscow, Russia